CLINICAL TRIAL: NCT01985828
Title: Prospective Evaluation of CyberKnife® as Monotherapy or Boost Stereotactic Body Radiotherapy for Intermediate or High Risk Localized Prostate Cancer
Brief Title: CyberKnife® as Monotherapy or Boost SBRT for Intermediate or High Risk Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5307
Record Dates: First submitted 2013-04-12; First posted 2013-11-15 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: Prostate Adenocarcinoma
Keywords: Prostate neoplasm; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Androgen Antagonists; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intermediate Risk (Experimental): Short term (4-6 months) androgen deprivation therapy (ADT) per current standard of care + CyberKnife 21 Gy (7 Gy x 3) and Prostate/SV Intensity Modulated radiation therapy (IMRT) 45-50.4 Gy
  OR
  Short term (4-6 months)androgen deprivation therapy + CyberKnife 36.35 Gray (7.27 Gray x 5)
  Interventions: Radiation: CyberKnife; Other: Androgen Deprivation Therapy (ADT); Radiation: Intensity Modulated radiation therapy (IMRT)
- High Risk (Experimental): Short or Long term (6 months - 3 years) androgen deprivation therapy (ADT) + 45-50.4 Gy and Pelvis Intensity Modulated radiation therapy (IMRT) per current standard of care + 21 Gy (7 Gy x 3) CyberKnife boost
  Interventions: Radiation: CyberKnife; Other: Androgen Deprivation Therapy (ADT); Radiation: Intensity Modulated radiation therapy (IMRT)

INTERVENTIONS:
Radiation: CyberKnife
Other: Androgen Deprivation Therapy (ADT)
Radiation: Intensity Modulated radiation therapy (IMRT) — Per current standard of care

SUMMARY:
The primary objective of this study is to document the effectiveness of Cyberknife stereotactic body radiotherapy (SBRT) in the treatment of intermediate and high-risk localized prostate cancer defined by biochemical Disease-Free Survival (bDFS), using Phoenix and American Society of Therapeutic Radiation and Oncology (ASTRO) definitions, at 5 years.

During the prostate-specific antigen era, an ever-increasing percentage of men with prostate cancer have presented with clinically localized, potentially curable disease. Although conventional treatment options are potentially curative in selected patients, these treatments also have drawbacks, including the risk of negative long-term quality of life consequences and serious complications.

The CyberKnife® system is a type of radiation machine that uses a special system to precisely focus large doses of x-rays on the tumor. The device is designed to concentrate large doses of radiation onto the tumor so that injury from radiation to the nearby normal tissue will be minimal.

Intermediate risk patients will be treated with either CyberKnife® Stereotactic Body Radiation Therapy (SBRT) monotherapy or CyberKnife® SBRT boost followed by Intensity Modulated Radiation Therapy (IMRT). High risk patients will be treated with CyberKnife® SBRT boost followed by IMRT. Treatment will last 4-7 days. Patients will complete the QOL questionnaires before treatment. Questionnaires will also be completed during follow-up visits at 1, 3 , 6, 12, 18, 24, 30 and 36 months then every 12 months until year 5.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate the efficacy and Health-Related Quality of Life (HRQOL) in intermediate and high-risk prostate cancer patients treated with SBRT as monotherapy or as a boost in combination with IMRT.

ELIGIBILITY:
* Patient must be ≥ 18 years of age.
* Histologically proven prostate adenocarcinoma

  * Gleason score 2-10 (reviewed by reference lab)
  * Biopsy within one year of date of registration
  * Clinical stage T1b-T4, N0-Nx, M0-Mx (AJCC 7th Edition)
  * T-stage and N-stage determined by physical exam and available imaging studies (ultrasound, CT, and/or MRI; see section 4.5)
  * M-stage determined by physical exam, CT or MRI. Bone scan not required unless clinical findings suggest possible osseous metastases.
* PSA ≤ 50 ng/ml, CBC, platelets, BUN, creatinine prior to treatment
* Patients belonging in one of the following risk groups:

  * Intermediate: CS T2b-c and Gleason <6 and PSA ≤ 10, or CS T1b-T2b, and Gleason 7 and PSA ≤ 10 ng/ml, or Gleason <6 and PSA 11-20 ng/ml
  * High: CS T3-4, Gleason score >7and PSA<50
* Prostate volume: ≤ 100 cc

  * Determined using: volume = π/6 x length x height x width
  * Measurement from MRI, CT or ultrasound prior to registration.
* ECOG performance status 0-1
* No prior prostatectomy or cryotherapy of the prostate
* No prior radiotherapy to the prostate or lower pelvis
* No implanted hardware or other material that would prohibit appropriate treatment planning or treatment delivery, in the investigator's opinion.
* No chemotherapy for a malignancy in the last 5 years.
* No history of an invasive malignancy (other than this prostate cancer, or basal or squamous skin cancers) in the last 5 years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arica Hirsch, MD, Principal Investigator — Advocate Lutheran General Hospital; Majid M Mohiuddin, MD, Study Chair — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intermediate Risk: Short term (4-6 months) androgen deprivation therapy (ADT) per current standard of care + CyberKnife 21 Gy (7 Gy x 3) and Prostate/SV Intensity Modulated radiation therapy (IMRT) 45-50.4 Gy
  OR
  Short term (4-6 months)androgen deprivation therapy + CyberKnife 36.35 Gray (7.27 Gray x 5)
  CyberKnife
  Androgen Deprivation Therapy (ADT)
  Intensity Modulated radiation therapy (IMRT): Per current standard of care
- High Risk: Short or Long term (6 months - 3 years) androgen deprivation therapy (ADT) + 45-50.4 Gy and Pelvis Intensity Modulated radiation therapy (IMRT) per current standard of care + 21 Gy (7 Gy x 3) CyberKnife boost
  CyberKnife
  Androgen Deprivation Therapy (ADT)
  Intensity Modulated radiation therapy (IMRT): Per current standard of care
Period: Overall Study
Arm/Group | Intermediate Risk | High Risk
Started | 53 | 30
Completed | 47 | 29
Not Completed | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermediate Risk | High Risk | Total
Number analyzed (Participants) | 53 | 30 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 39 | 19 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 53 | 30 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 30 | 83

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Disease-Free Survival (bDFS), Using Phoenix and ASTRO Definitions
Description: Phoenix definition: Biochemical recurrence of prostate cancer (PCa) after curative radiotherapy defined as a prostate-specific antigen (PSA) rise of ≥2 ng/ml above the nadir.
  Astro definition: Biochemical failure in prostate cancer defined as three consecutive rises in prostate-specific antigen (PSA) after a nadir.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk | High Risk
Number analyzed (Participants) | 47 | 29
Participants
  Phoenix Definition | 46 | 27
  Astro Definition | 45 | 27

2. Secondary Outcome: Measure the Rates of Acute and Late Grade 3-5 Gastrointestinal and Genitourinary Toxicity
Description: Acute toxicity is graded based upon Common Terminology Criteria for Adverse Events (CTCAE). The Common Terminology Criteria for Adverse Events (CTCAE) v3.0 is a standardized system used to classify and grade the severity of adverse events (AEs) experienced by cancer patients during treatment, with a grading scale ranging from 1 (mild) to 5 (death).
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intermediate Risk | High Risk
Number analyzed (Participants) | 47 | 29
Participants | 2 | 5

3. Secondary Outcome: Expanded Prostate Cancer Index Composite Epic-26
Description: The 26-item version of EPIC, also known as EPIC Short Form or EPIC-26, contains five symptom domains (urinary incontinence, urinary irritative/obstructive, sexual, bowel, hormonal), scored from 0 (worst) to 100 (best).
Time Frame: 3 years
Measure: Least Squares Mean (Full Range); unit: units on a scale
Arm/Group | Intermediate Risk | High Risk
Number analyzed (Participants) | 47 | 29
units on a scale | 78.73 [37.88 to 95.60] | 78.73 [37.88 to 95.60]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Intermediate Risk | High Risk
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/30
Other Adverse Events (participants affected / at risk) | 0/53 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT01985828/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-18): https://cdn.clinicaltrials.gov/large-docs/28/NCT01985828/ICF_001.pdf